CLINICAL TRIAL: NCT04739592
Title: The Effect of Alendronate Sodium Vitamin D3 Tablets on Knee Joint Structure and Knee Osteoarthritis Pain: A Multi-center, Randomized, Double-blind, Controlled Study.
Brief Title: A Study of Alendronate Sodium Vitamin D3 Tablets on Knee Osteoarthritis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Peking UMCH
Record Dates: First submitted 2021-01-13; First posted 2021-02-04 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2021-09

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- alendronate sodium vitamin D3 tablets (Experimental): participants will receive alendronate sodium vitamin D3 tablets once per week for one year.
  Interventions: Drug: alendronate sodium vitamin D3 tablets
- placebo (Placebo Comparator): participants will receive a placebo tablet once per week for one year.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: alendronate sodium vitamin D3 tablets — once per week for one year
  Arms: alendronate sodium vitamin D3 tablets
Drug: Placebo — once per week for one year
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effect of alendronate sodium vitamin D3 tablets compared with placebo on the improvement of joint structure and joint pain in participants with knee osteoarthritis. The treatment period of this study is one year and followed-up period is 2 years. The results of knee joint MRI will be evaluated by using the WORMS score.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double-blind, placebo-controlled study This study is planned to commence after obtaining Ethics Committee approval. participants will be randomised to a one-year course of alendronate sodium vitamin D3 tablets or placebo. 1:1 double blinded randomisation will be undertaken. This study plans to enroll 60 participants and will be carried out in three domestic centers (Peking Union Medical College Hospital, Zhongshan Hospital and The Third Affiliated Hospital of Southern Medical University) with a follow-up period of 2 years.

As the main goal of this exploratory study is to evaluate the effect of alendronate sodium vitamin D3 tablets compared with placebo on the improvement of joint structure and joint pain in participants with knee osteoarthritis. The primary outcome measure is WORMS score of knee joint MRI at 6 months and 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with significant knee pain (pain score≥40mm on the 100mmVAS scale);
2. Male or female patients, between 50-75 years old;
3. MRI suggests bone marrow edema-like lesions;
4. Knee osteoarthritis (in accordance with the diagnostic criteria of American College of Rheumatology (ACR) and Chinese Orthopaedic Association);
5. Kellgren-Lawrence gradingⅠorⅡin X-ray;

Exclusion Criteria:

1. Other forms of active arthritis (such as rheumatoid arthritis or other inflammatory arthritis);
2. Taken non-steroidal anti-inflammatory drugs and central analgesics (such as opioids) within two weeks；
3. Liver function ALT or AST is 1.5 times the upper limit of normal； creatinine clearance <35ml/min；
4. Pregnancy or suckling;
5. Serious heart disease, endocrine, digestive, mental, nervous system diseases or cancer;
6. Active ulcers and a history of upper gastrointestinal bleeding;
7. Esophageal motility disorders, such as esophageal tardiness or stenosis;
8. Renal dysfunction or osteomalacia;
9. Tobacco addiction (mean 10 cigarettes per day or more) or/and alcohol addiction (mean 50ml per day or more);
10. Fresh fracture in the last six months;
11. Serious illnesses and life expectancy<2 years;
12. Allergic to study drugs;
13. Used any study drug or device within 30 days before randomization or within the drug half-life (whichever is longer);
14. Failure to take medication as required;
15. Replacement surgery in the near future;
16. Contraindications to MRI scans (e.g. implanted pacemakers, metal sutures, shrapnel or iron filings in the eyes, claustrophobia, knees too large to use coils);
17. Sensitive to or unsuitable for X-ray exposure (e.g. aplastic anemia, etc);
18. Poor dental health or dental surgery in the near future.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-07 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
WORMS score of knee joint MRI | The sixth month
  WORM score of participants at the sixth month after enrollment
WORMS score of knee joint MRI | The 12th month
  WORM score of participants at the 12th month after enrollment

SECONDARY OUTCOMES:
WORMS score of knee joint MRI | The 24th month
  WORM score of patients at the 24th month after enrollment
Pain intensity and symptom record | The second week
  Pain intensity and symptom record of patients at the second week after enrollment
Pain intensity and symptom record | The 4th week
  Pain intensity and symptom record of patients at the 4th week after enrollment
Pain intensity and symptom record | The 8th week
  Pain intensity and symptom record of patients at the 8th week after enrollment
Pain intensity and symptom record | The 12th week
  Pain intensity and symptom record of patients at the 12th week after enrollment
Quality of life (the MOS item short from health survey,SF-36 ) | The third month
  SF-36 scale of patients at the third month after enrollment
Quality of life (the MOS item short from health survey,SF-36 ) | The sixth month
  SF-36 scale of patients at the sixth month after enrollment. The score is calculated from eight dimensions, with the higher the final score the better
Quality of life (the MOS item short from health survey,SF-36 ) | The 12th month
  SF-36 scale of patients at the 12th month after enrollment. The score is calculated from eight dimensions, with the higher the final score the better
bone density (lumbar spine, hip joint and knee joint) | The 12th month
  bone density of patients at the 12th month after enrollment
bone density (lumbar spine, hip joint and knee joint) | The 24th month
  bone density of patients at the 24th month after enrollment
Risk of knee replacement | The 12th month
  Risk of knee replacement of patients at the 12th month after enrollment
Risk of knee replacement | The 24th month
  Risk of knee replacement of patients at the 24th month after enrollment
Kellgren & Lawrence(KL) grading Score | The 12th month
  KL-grading Score of patients at the 12th month after enrollment, 0 to Ⅳ, higher scores mean a worse outcome
Kellgren & Lawrence(KL) grading Score | The 24th month
  KL-grading Score of patients at the 12th month after enrollment, 0 to Ⅳ, higher scores mean a worse outcome
Serum IL-6, TNF-a, erythrocyte sedimentation rate, C-reactive protein | The third month
  Serum inflammatory factor of patients at the third month after enrollment, IL-6 and TNF-a were measured in pg/ml,erythrocyte sedimentation rate was measured in mm/h, C-reactive protein was measured in mg/dL.
Serum IL-6, TNF-a, erythrocyte sedimentation rate, C-reactive protein | The sixth month
  Serum inflammatory factor of patients at the sixth month after enrollment, IL-6 and TNF-a were measured in pg/ml,erythrocyte sedimentation rate was measured in mm/h, C-reactive protein was measured in mg/dL.
Serum IL-6, TNF-a, erythrocyte sedimentation rate, C-reactive protein | The 12th month
  Serum inflammatory factor of patients at the 12th month after enrollment, IL-6 and TNF-a were measured in pg/ml,erythrocyte sedimentation rate was measured in mm/h, C-reactive protein was measured in mg/dL.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Peking Union Medical College Hospital, Beijing
  - The Third Affiliated Hospital of Southern Medical University, Guangzhou
  - Zhongshan Hospital, Shanghai

REFERENCES:
- [Derived] Peng HM, Weng XS, Li Y, Feng B, Qian W, Cai DZ, Zhao C, Yao ZJ, Yang Y, Zhang C, Wan S. Effect of alendronate sodium plus vitamin D3 tablets on knee joint structure and osteoarthritis pain: a multi-center, randomized, double-blind, placebo-controlled study protocol. BMC Musculoskelet Disord. 2022 Jun 17;23(1):584. doi: 10.1186/s12891-022-05521-4. PMID 35715774